CLINICAL TRIAL: NCT00551226
Title: Follow up of Autoantibodies in Active Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: 314-07
Record Dates: First submitted 2007-10-27; First posted 2007-10-30 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Tuberculosis
Keywords: TB; Patients with tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum of patients
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with tuberculosis
- 2: Healthy controls

SUMMARY:
We have previoulsy shown that patients with active Tuberculosis develop a wide array of autoantibodies including rheumatoid factor, anti-CCP, Antinuclear facyor and anti Sm antibodies. The purpose of this study is to evaluate whether the level of autoantibodies decrease after treatment aganist tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Active Tuberculosis treated

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with active tuberculosis who are currently receiving anti tuberculosis drugs
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-11; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Follow up after levels of autoantibodies | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ori Elkayam, M.D, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Tel Aviv, Israel